CLINICAL TRIAL: NCT03207412
Title: Clinical Study of Minimally Invasive Implantation of Human Amniotic Epithelial Cells in the Treatment of Premature Ovarian Insufficiency
Brief Title: Human Amniotic Epithelial Cells Treatment for Ovarian Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POI-2017
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive implantation (Experimental): Patients receive minimally invasive implantation, and 200 million hAECs is implanted into bilateral ovarian tissue by Ultrasound-guided puncture.
  Interventions: Biological: hAECs; Procedure: Minimally invasive implantation
- Intravenous infusion (Experimental): 100 million hAECs is administered by intravenous infusion every 30 days, for 3 times.
  Interventions: Biological: hAECs

INTERVENTIONS:
Biological: hAECs — human amniotic epithelial cells
Procedure: Minimally invasive implantation — Minimally invasive implantation with ultrasound guidance
  Arms: Minimally invasive implantation

SUMMARY:
This project will investigate the safety and effectiveness of human amniotic epithelial cells in primary ovarian insufficiency patients and provide a new cell therapy against infertility.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) refers to women before the 40 years of age who suffer clinical manifestations of ovarian recession. Now, there is no exact and effective treatment to restore ovarian function. Human amniotic Epithelial cells (hAECs) are derived from human amniotic epithelium. hAECs retain the characteristics of embryonic stem cells, as well as a strong differentiation potential and plasticity. Experiments show that the fertility of mice is significantly improved after amniotic epithelial cells implantation. In order to further study the role of hAECs in POI treatment, this project will conduct minimally invasive implantation with hAECs in 20 cases of POI patients, and evaluate the changes of ovarian function and the safety of hAECs implantation. hAECs is prepared by Chongqing iCELL Biotechnology Co.,Ltd., which is a subsidiary of Shanghai iCELL Biotechnology Co.,Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of POI, excluding genetic disease caused by patients; POI diagnostic criteria: Patients that <40 years of age, oligomenorrhea for 4 months,FSH> 25 IU/L.
2. Have fertility requirements;
3. Agree to sign the designed consent for the study.

Exclusion Criteria:

1. Breast cancer, ovarian cancer and other cancer/tumor;
2. Contraindications for pregnancy;
3. Coagulation disorder and other abnormal physical conditions.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2017-12-22 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of follicle stimulating hormone(FSH) | 1 year
  Serum FSH level is evaluated once a month after treatment.
antral follicle count (AFC) | 1 year
  the number of primordial egg follicles within the ovary per menstrual cycle

SECONDARY OUTCOMES:
Menstrual situation | 1 year
  Changes of menstrual cycle and menstrual period before and after treatment.
Luteinizing Hormone(LH) | 1 year
  serum level of LH
estrogen 2(E2) | 1 year
  serum level of E2
Anti Mullerian Hormone(AMH) | 1 year
  serum level of AMH
Ovarian volume | 1 year
  The ovarian volume is recorded by transvaginal ultrasound scan.

CONTACTS AND LOCATIONS:
Overall Officials: Chanyu Zhang, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: No